CLINICAL TRIAL: NCT03645746
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of Intravenously or Subcutaneously Administered REGN5069 in Healthy Volunteers
Brief Title: Safety, Tolerability, and Pharmacokinetics of REGN5069 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: R5069-HV-1810; 2018-000651-41 (EudraCT Number)
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Experimental): Cohort 1 will receive a single IV dose of REGN5069 or matching placebo
  Interventions: Drug: REGN5069; Drug: Placebo
- Cohort 2 (Experimental): Cohort 2 will receive a single sequential ascending IV dose of REGN5069 or matching placebo
  Interventions: Drug: REGN5069; Drug: Placebo
- Cohort 3 (Experimental): Cohort 3 will receive a single sequential ascending IV dose of REGN5069 or matching placebo
  Interventions: Drug: REGN5069; Drug: Placebo
- Cohort 4 (Experimental): Cohort 4 will receive a single sequential ascending IV dose of REGN5069 or matching placebo
  Interventions: Drug: REGN5069; Drug: Placebo
- Cohort 5 (Experimental): Cohort 5 will receive a single SC dose of REGN5069 or matching placebo
  Interventions: Drug: REGN5069; Drug: Placebo
- Cohort 6 (Experimental): Cohort 6 will receive a single sequential ascending SC dose of REGN5069 or matching placebo
  Interventions: Drug: REGN5069; Drug: Placebo
- Cohort 7 (Experimental): Cohort 7 will receive a single sequential ascending IV dose of REGN5069 or matching placebo
  Interventions: Drug: REGN5069; Drug: Placebo

INTERVENTIONS:
Drug: REGN5069 — REGN5069 will be administered by IV infusion or SC injection
Drug: Placebo — Placebo-matching REGN5069

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of single ascending doses of REGN5069 administered intravenously (IV) and subcutaneously (SC) in healthy male and female participants.

The secondary objectives of the study are to characterize the pharmacokinetics (PK) profile of single IV and SC doses of REGN5069 in healthy participants and assess the immunogenicity of REGN5069 in healthy participants administered single IV or SC doses of REGN5069

ELIGIBILITY:
Key Inclusion Criteria:

* Participant is judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, and ECG performed at screening and/or prior to study drug dosing
* Participant is in good health based on laboratory safety testing obtained at the screening visit
* Willing and able to comply with clinic visits and study-related procedures
* Provide informed consent signed by study participant or legally acceptable representative

Key Exclusion Criteria:

* History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric or neurological disease
* Has any physical examination findings and/or history of any illness that might confound the results of the study or poses an additional risk to the subject by study participation
* Hospitalization for any reason within 60 days of the screening visit
* Current cigarette smoker or former smoker (cigarettes or e-cigarettes) who stopped smoking within 3 months prior to screening
* History of drug or alcohol abuse within a year prior to the screening visit
* Presence of HIV, hepatitis B, or hepatitis C seropositivity at screening or within 3 months prior to dosing with the exception of false positive screening tests as documented by polymerase chain reaction or Western blot
* Any malignancy within the past 5 years, except for basal cell or squamous epithelial cell carcinomas of the skin or carcinoma in situ of the cervix or anus, that have been resected, with no evidence of metastatic disease for 3 years

Note: Other protocol Inclusion/Exclusion Criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | From baseline up to week 36
Incidence of laboratory abnormalities | From baseline up to week 36
  As measured by chemistry, hematology and urinalysis
Incidence of vital signs abnormalties | From baseline up to week 36
  As measured by heart rate, blood pressure, body temperature and respiratory rate
Incidence of standard 12-lead electrocardiogram (ECG) abnormalties | From baseline up to week 36
  As measured by heart rate, PR, complex of Q, R, and S waves [QRS], QT-intervals, and QTc

SECONDARY OUTCOMES:
Concentration of REGN5069 in serum over time | From baseline up to week 36
Incidence of anti-drug antibody (ADA) | From baseline up to week 36

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Research Facility, Ghent, Belgium